CLINICAL TRIAL: NCT00382837
Title: A Phase III Multi-Center, OpenLabel, Follow-Up Study to Assess the Safety & Efficacy of Epratuzumab in Patients With Acute Severe SLE Flares Excluding the Renal or Neurologic Systems
Brief Title: Study of Epratuzumab in Systemic Lupus Erythematosus
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SL0005; EudraCT# 2006-003865-15
Record Dates: First submitted 2006-09-29; First posted 2006-10-02 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2007-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus,; Antibody,; B-Cell immunotherapy
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — epratuzumab

INTERVENTIONS:
Drug: Epratuzumab

SUMMARY:
Epratuzumab is an investigational antibody designed to help treat SLE. The purpose is to evaluate safety and long term efficacy in concert with standard SLE treatments

ELIGIBILITY:
Inclusion Criteria:

* Must have completed SL0003 Alleviate A through 48 weeks

Exclusion Criteria:

* Development of toxicity to Epratuzumab
* Significant protocol deviations from SL0003 Study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01

PRIMARY OUTCOMES:
The primary objective is to continue to gather long term safety data on patients with moderate to severe flaring SLE.

SECONDARY OUTCOMES:
To continue to assess the efficacy and tolerability of epratuzumab;
To continue to monitor the plasma concentration and immunogenicity profile of epratuzumab in patients with Lupus;
To continue to assess epratuzumab on Health-related quality of life in lupus patients;
To continue to assess disease status as reported by the patient and physician.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Barry, Study Director — UCB Pharma
Locations (54):
- United States (20):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Los Angeles, California
  - Upland, California
  - Farmington, Connecticut
  - Washington D.C., District of Columbia
  - Aventura, Florida
  - Chicago, Illinois
  - Baltimore, Maryland
  - New York, New York
  - Syracuse, New York
  - The Bronx, New York
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Gallipolis, Ohio
  - Tulsa, Oklahoma
  - Charleston, South Carolina
  - Dallas, Texas
  - Arlington, Virginia
  - Edmonds, Washington
- Belgium (2):
  - Brussels
  - Liège
- Brazil (4):
  - Rio de Janeiro, Rio de Janeiro
  - Goiânia
  - Rio de Janeiro
  - São Paulo
- Winnipeg, Manitoba, Canada
- Czechia (3):
  - Hradec Králové
  - Olomouc
  - Prague
- France (2):
  - Paris
  - Toulouse
- Germany (4):
  - Erlangen
  - Heidelberg
  - Mannheim
  - München
- Hungary (2):
  - Debrecen
  - Pécs
- Italy (2):
  - Ancona
  - Brescia
- Netherlands (3):
  - Amsterdam
  - Groningen
  - Leiden
- Piešťany, Slovakia
- Spain (4):
  - Barcelona
  - Madrid
  - Santander
  - Seville
- United Kingdom (6):
  - Leeds, West Yorkshire
  - Birmingham
  - London
  - Manchester
  - Newcastle upon Tyne
  - Sheffield